CLINICAL TRIAL: NCT01479712
Title: Intra-abdominal at Cesarean Section: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM11572
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Nausea; Vomiting
Keywords: Irrigation; Cesarean Section; Nausea; Infection
MeSH Terms: conditions — Nausea; Vomiting; Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irrigation (Active Comparator): This is the arm that will receive irrigation.
  Interventions: Procedure: Normal Saline Irrigation
- No Irrigation (No Intervention): This is the arm that will not receive irrigation.

INTERVENTIONS:
Procedure: Normal Saline Irrigation — Irrigation with warm normal saline into the abdominal cavity. Approximately 500-1000cc.
  Arms: Irrigation

SUMMARY:
The purpose of this study is to determine if intra-abdominal irrigation at the time of cesarean delivery increased maternal GI discomfort without affecting infection rates.

We hypothesized that avoiding intra-operative irrigation at the time of cesarean delivery will decrease intra-operative nausea and vomiting without increasing maternal infectious morbidity, post-operative pain, return of bowel function, or time to discharge.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled trial.

Based on available literature and clinical experience, we expect a twenty percent decrease in gastrointestinal disturbances by avoiding intraoperative irrigation at the time of cesarean section. With the type 1 error rate set at 0.05 and a power of 0.90; this will require 184 patients in each arm (irrigation versus no irrigation) to obtain an adequate sample size. Paper copies of written consent and any identifying information will be kept in a secured, locked file. All data collected will be stored in a password protected computer file that will be accessible only to the investigators.

Patients will be identified at the time of admission to the Labor and Delivery unit. A physician will discuss the study with the patient. After time for consideration and having had all questions answered the patient will then be consented for the trial. Consent will be obtained at the time of admission to the Labor and Delivery unit. If the patient has a successful vaginal delivery the patient will not enter the study. If the patient requires a cesarean section the patient will be randomized either in to an irrigation or a nonirrigation group. Assignment will be performed by pulling sequentially numbered opaque envelopes containing computer-randomized individual allocations. This randomization will be carried out by research staff before the initiation of the study, and the patients will be blinded to treatment once assigned. Information regarding basic demographic data, comorbidities that may affect infection rates (diabetes, hypertension, ect), interventions during labor, and post partum course will be obtained from the patients' charts.

The two arms will differ only in intraoperative management of the patient after delivery of the baby. Patients in the irrigation arm will receive a cesarean section with irrigation of the abdominal cavity with 500-1000mL of warm normal saline after closure of the uterine incision but prior to the closure of the abdominal wall. In addition all blood clots and other debris will be evacuated from the paracolic gutters, anterior and posterior culdesacs, and under the bladder flap. The nonirrigation group will receive Joel-Cohen cesarean section without the irrigation with normal saline. This group will also have any large debris including blood clots evacuated. Both groups will undergo standard closure of the abdominal wall, including reapproximation of the rectus muscles and suturing of the rectus fascia with running nonlocking absorbable suture. Prefascial irrigation of the subcutaneous tissues superior to the closed fascia will be done in both groups. Staples or absorbable suture will be used for skin closure. In addition all patients will receive a standardized dose of 1 gram of a first generation cephalosporin or 900mg clindamycin intravenously as antibiotic prophylaxis at the time of umbilical cord clamping.

As per standard of care, the post partum care will include vital signs every 4 hours including patient report of pain level and nausea, discontinuation of the foley catheter and advancement of the diet on postoperative day one, daily examination of the incision, notation of return of gastrointestinal function, early ambulation, and a complete blood count on the first postoperative day.

The primary outcome of measure will be maternal GI disturbance. This will be defined as nausea or emesis during the cesarean section as well as any nausea requiring medical intervention during her hospitalization. The time to return of bowel function will also be recorded. The secondary outcome of measure is the incidence of maternal infectious morbidity, defined as endometritis. This will be diagnosed with two or more of the following are present: abnormally tender uterus on exam, temperature greater than 100.4°F at any time postoperatively, unexplained maternal tachycardia greater than 100 beats per minute. Patients will also be monitored for wound infections daily by visual inspection of the incision. Diagnosis will be made if any erythema, tenderness, discharge or separation occurs with maternal fever. Post operative care providers will be blinded to group assignment to avoid any potential bias.

The investigators will collect the data, perform data entry, and review charts to ensure accuracy of information provided by the treating physician. Periodic reviews of the data entry will be performed to ensure completeness and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* 18 years of age or older
* presenting to MCV Hospital
* undergoing obstetrically indicated cesarean section
* english speaking

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Intra-operative nausea | intra-operative
  Any nausea reported by the patient during the cesarean section

SECONDARY OUTCOMES:
Post operative GI disturbance | 2-3 days post operatively
  Any nausea or vomiting reported or observed during the patient's postoperative period
Infection | 2-3 days post operatively
  Any documented infection during the patient's postoperative stay

CONTACTS AND LOCATIONS:
Overall Officials: Christine Isaacs, MD, Principal Investigator — VCU Department of Obstetrics and Gynecology
Locations (1):
- Virginia Commonwealth University Hospital System, Richmond, Virginia, United States

REFERENCES:
- [Derived] Viney R, Isaacs C, Chelmow D. Intra-abdominal irrigation at cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2012 Jun;119(6):1106-11. doi: 10.1097/AOG.0b013e3182460d09. PMID 22617574